CLINICAL TRIAL: NCT01978548
Title: A Double-blind, Placebo-Controlled, Randomized, 4-Week, Multiple-Dose, Proof-of-Mechanism Study in Subjects With Prodromal Alzheimer's Disease Investigating the Effects of JNJ-54861911 on Aβ Processing in CSF and Plasma
Brief Title: A Study to Evaluate the Effects of JNJ-54861911 on Amyloid Beta Processing in Cerebrospinal Fluid and Plasma in Patients With Prodromal Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103012; 54861911ALZ1005 (Other: Janssen Research & Development, LLC); 2013-003036-69 (EudraCT Number)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Prodromal Alzheimer Disease; Safety; Tolerability; Pharmacokinetic; Proof of Mechanism; JNJ-54861911
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- JNJ-54861911 10 mg (Experimental): From Day 1 to Day 28 inclusive, patients will self-administer once daily study drug (JNJ-54861911 or placebo) with a glass of non-carbonated water (approximately 200 mL).
  Interventions: Drug: JNJ-54861911 10 mg
- JNJ-54861911 50 mg (Experimental)
  Interventions: Drug: JNJ-54861911 50 mg
- Placebo (Placebo Comparator): Patients will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-54861911 10 mg — JNJ-54861911 10 mg will be administered as two 5 mg oral tablets once daily.
  Arms: JNJ-54861911 10 mg
Drug: JNJ-54861911 50 mg — JNJ-54861911 50 mg will be administered as two 25 mg oral tablets once daily.
  Arms: JNJ-54861911 50 mg
Drug: Placebo — Matching placebo will be administered as 2 oral tablets once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of JNJ-54861911 in patients with prodromal Alzheimer's disease (pAD).

DETAILED DESCRIPTION:
This will be a multicenter, double-blind (neither investigator nor patient knows which treatment the patient receives), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), randomized (patients are assigned different treatments based on chance), multiple-dose, proof-of-mechanism (POM) study in pAD. Approximately 24 outpatients (n=8/treatment group) diagnosed with pAD, according to the inclusion and exclusion criteria, will participate in this 4-week treatment study. For all enrolled patients, this study will consist of an 8-week eligibility screening period, a 4-week double-blind treatment period, and a follow-up examination (7-14 days after the last dose). Patients will be assigned randomly to 1 of 3 treatment groups: placebo, JNJ-54861911 10 mg once daily, or JNJ-54861911 50 mg once daily. Safety assessments will be performed throughout the study. The maximal study duration for a patient will be 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had sufficient education or work experience to exclude mental retardation
* Patients must have an abnormal cognitive performance consistent with mild cognitive impairment based on the computerized neuropsychological test battery (CANTAB Elect) that can effectively screen patients and identify cognitive deficits consistent with mild cognitive impairment
* Patients must have evidence of amyloid deposition by means of either 1) low cerebrospinal fluid amyloid beta 1-42 (CSF amyloid beta 1-42) levels and elevated CSF p-Tau and/or total tau levels at screening (cut off values for CSF amyloid beta 1-42 and CSF p-tau and/or total tau will be based on the values established by the Clinical Neurochemistry Lab, Sahlgrenska University Hospital, Mölndal, Sweden and specified in a separate lab manual) or 2) a positive 18F-flutematol amyloid positron emission tomography (PET) amyloid scan at screening (optional depending on the site's PET capability) or both
* Patients must have a body mass index (BMI=weight/height²) between 18 and 35 kg/m2, inclusive, at screening
* Women must be postmenopausal, permanently sterilized or otherwise be incapable of pregnancy
* Must adhere to required contraception during and for 3 months after study
* Patients must be otherwise healthy for their age group or medically stable with or without medication
* Patients must be able to be compliant with self-administration of medication
* Patients must be able to swallow drug as a whole

Exclusion Criteria:

* Patient has evidence of brain disease, other than Alzheimer's Disease (AD), or any other abnormality (e.g. folic acid/Vitamin B12 deficiency) that could explain the cognitive deficit (including, but not limited to vascular encephalopathy or strokes, as imaged by cerebral MRI and Major Depression, as defined by DSM-IV criteria)
* Patient has been diagnosed with dementia due to AD, due to other diseases, or with AD and contribution of other disorders (mixed dementia)
* Patient has evidence of familial autosomal dominant AD
* Patient has a history of substance or alcohol abuse
* Relevant history of lower back pain or scoliosis and/or major (lumbar) back surgery
* Patient is allergic to local anesthetics and/or iodine or chlorhexidine
* Patient has taken aspirin (even low dose) within 5 days prior to lumbar puncture (screening or Day 1)
* Patient has taken Low Molecular Weight Heparin (LMWH) within 12 hours prior to lumbar puncture (screening or Day 1)
* Patient has taken any anticoagulant treatment (e.g. warfarin; besides LMWH described above) within 1 week prior to lumbar puncture (screening or Day 1)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Levels of amyloid beta 1-40 in cerebrospinal (CSF) after treatment at the intended target dose range | Up to 4 weeks
Levels of amyloid beta 1-40 in plasma after treatment at the intended target dose range | Up to 4 weeks
Maximum observed plasma concentration (Cmax) of JNJ-54861911 | Up to 4 weeks
  Cmax is the observed maximum plasma concentration of study drug, taken directly from the plasma concentration-time profile
Time to reach maximum observed plasma concentration of JNJ-54861911 | Up to 4 weeks
  Time when Cmax is observed, taken directly from the plasma concentration-time profile
Area under the plasma concentration time curve (AUC) from 0 to t hours of JNJ-54861911 | Up to 4 weeks
  Area under the plasma concentration-time curve from 0 to t hours post dosing (time t is the dosing interval)
Half-life of JNJ-54861911 | Up to 4 weeks
  Elimination half-life associated with the terminal slope of the semi-logarithmic drug concentration-time curve, calculated as 0.693/terminal slope
Cerebrospinal fluid exposure of JNJ-54861911 | Up to 4 weeks
The number of volunteers who experience adverse events as a measure of safety and tolerability of JNJ-54861911 after multiple-dose administration in the anticipated target dose range | Up to 4 weeks

SECONDARY OUTCOMES:
Levels of amyloid beta fragments (amyloid beta 1-37, 1-38, and 1-42) in cerebrospinal fluid after treatment at the intended target dose range | Up to 4 weeks
Levels of amyloid beta fragments (amyloid beta 1-37, 1-38, and 1-42) in plasma after treatment at the intended target dose range | Up to 4 weeks
Levels of amyloid precursor protein (APP) fragments (soluble amyloid precursor protein α [sAPPalpha], sAPPbeta, totalAPP) in CSF after treatment at the intended target dose range | Up to 4 weeks
Compare the relationship of amyloid beta 1-40 levels in plasma and cerebrospinal fluid after treatment at the intended target dose range | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- Belgium (3):
  - Antwerp
  - Ghent
  - Hoboken
- Amsterdam, Netherlands
- Spain (4):
  - Barcelona
  - Madrid
  - Terrassa
  - Valencia
- Sweden (2):
  - Mölndal
  - Stockholm

REFERENCES:
- [Derived] Timmers M, Streffer JR, Russu A, Tominaga Y, Shimizu H, Shiraishi A, Tatikola K, Smekens P, Borjesson-Hanson A, Andreasen N, Matias-Guiu J, Baquero M, Boada M, Tesseur I, Tritsmans L, Van Nueten L, Engelborghs S. Pharmacodynamics of atabecestat (JNJ-54861911), an oral BACE1 inhibitor in patients with early Alzheimer's disease: randomized, double-blind, placebo-controlled study. Alzheimers Res Ther. 2018 Aug 23;10(1):85. doi: 10.1186/s13195-018-0415-6. PMID 30134967